CLINICAL TRIAL: NCT04338425
Title: Patient Satisfaction With Postoperative Communication Modality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-01489
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Communication group (No Intervention): Participants will not communicate with their surgeons until the post operative office visit.
- Voice call group (Active Comparator): Participants will receive voice call from the surgeon after being discharged and before their post operative office visit.
  Interventions: Behavioral: Voice call
- Video call group (Active Comparator): Participants will receive video call from surgeon after being discharged and before their post operative office visit
  Interventions: Behavioral: Video call

INTERVENTIONS:
Behavioral: Voice call — Attending surgeons will contact with their patients on the day of surgery after discharge via voice call.
  Arms: Voice call group
Behavioral: Video call — Attending surgeons will contact with their patients on the day of surgery after discharge via video call (video conferencing application such as FaceTime or Skype)
  Arms: Video call group

SUMMARY:
Communication between a surgeon and a patient in the immediate postoperative period is thought to influence patient satisfaction. There is currently no standard of care regarding the optimal form of postoperative communication, nor is there a consensus in our department as to which modality is preferred by patients.The purpose of this study is to determine which form of communication, if any, is preferred by patients. Furthermore, this study aims to evaluate the impact that various forms of communication during the immediate postoperative period have on patient (subject) satisfaction. The study hypothesizes that patient (subject) satisfaction with their surgeon will be highest among those who communicate with their surgeons via videotelephony (i.e., videoconferencing) and that the lowest satisfaction will be among patients (subjects) who did not communicate with their surgeon until their regularly scheduled postoperative office visit. The results of this study may help identify low cost methods for increasing patient satisfaction.

DETAILED DESCRIPTION:
This is a prospective, randomized study designed to evaluate the effects of different communication modalities between surgeons and patients (subjects) in the immediate postoperative period. Given the nature of the study, it is not possible for either the surgeons or the subjects to be blinded. To reduce bias that may occur due to each surgeon's personal preference for postoperative communication modality, the surgeons (rather than individual subjects) will be randomized to one of the three communication modality groups (no communication on the day of surgery, voice call, or videoconferencing).

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery at the NYU Langone Orthopedic Center

Exclusion Criteria:

* Under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 295 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Percent of participants' satisfaction with surgeon | post operative office visit (1 week after surgery)
  The first self reported survey is designed specifically for this study to assess participants' satisfaction with their experience and postoperative communication.

SECONDARY OUTCOMES:
Percent of participants' satisfaction with hospital experience | post operative office visit (1 week after surgery)
  The second self reported survey contains questions from the standard HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) survey, which has been validated and used extensively to assess subject satisfaction with hospital experience.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and upon reasonable request. Requests should be directed to matthew.kingery@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.